CLINICAL TRIAL: NCT01599117
Title: Udenafil Therapy to Improve Symptomatology, Exercise Tolerance and Hemodynamics in Patients With Heart Failure With Preserved Ejection Fraction: Phase III, Randomized, Double-blind, Placebo-controlled Trial [ULTIMATE-HFpEF Trial]
Brief Title: A Randomized Trial of Udenafil Therapy in Patients With Heart Failure With Preserved Ejection Fraction [ULTIMATE-HFpEF]
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Yong-Jin Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1202-006-396
Record Dates: First submitted 2012-05-13; First posted 2012-05-15 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Diastolic Heart Failure
Keywords: Heart Failure with Preserved Ejection Fraction; Diastolic Heart Failure; Exercise Capacity; Cardiopulmonary Exercise Test; Udenafil (Zydena); Phosphodiesterase Type 5 Inhibitors
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo arm (Placebo Comparator): Capsule that is identically appearing with udenafil will be administered to patients in placebo group. For the first 4 weeks, patients will receive 50 mg of placebo drug two times a day, and then the dosage will be doubled to 100 mg two times a day for next 8 weeks.
  Interventions: Drug: Placebo
- Udenafil (Active Comparator): Patients will receive 50 mg of udenafil two times a day, and then the dosage will be doubled to 100 mg two times a day for next 8 weeks.
  Interventions: Drug: Udenafil (Zydena)

INTERVENTIONS:
Drug: Placebo — Capsule, appears identical with udenafil, will be provided by Dong-A pharmaceutical company. Patients will receive 50 mg of placebo drug two times a day for 4 weeks, and then the dosage will be escalated to 100 mg two times a day for next 8 weeks.
  Other Names: The same placebo drug of NCT01553721.
  Arms: Placebo arm
Drug: Udenafil (Zydena) — Udenafil (Zydena), a newly developed PDE-5 inhibitor by Dong-A pharmaceutical company, will be administered to patients in this group, 50 mg two times a day for 4 weeks, and then the dosage will be escalated to 100 mg two times a day for next 8 weeks.
  Other Names: DA-8159 (CAS No 268203-93-6)
  Arms: Udenafil

SUMMARY:
The investigators hypothesized that udenafil, a newly developed phosphodiesterase type 5 inhibitor, would improve symptom, exercise capacity and hemodynamic status in patients with heart failure with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) had been considered as a milder form of heart failure until 1990's. However, the prevalence and the prognosis of HFpEF were found to be similar to that of heart failure with reduced ejection fraction (HFrEF) and it is widely accepted that HFpEF is a separate entity of heart failure, substantially different from HFrEF. The pathophysiology of HFpEF can be contracted to the increased stiffness and impaired relaxation of left ventricle (LV), causing increased LV end-diastolic pressure and pulmonary venous pressure. These may lead to dyspnea, limited exercise capacity, and pulmonary congestion in patients.

Current guidelines on treatment of HFpEF include appropriate blood pressure control, rate control in those with atrial fibrillation, and use of diuretics for pulmonary or peripheral edema. But there has been no evidence-based effective treatment strategy for HFpEF. Recently, phosphodiesterase type 5 (PDE-5) inhibitors (eg. sildenafil, vardenafil, tadalafil) have shown promising effects on heart failure, reducing pulmonary vascular resistance, improving LV systolic and diastolic function, exercise capacity and quality of life. These results infer that PDE-5 inhibitors might be beneficial in patients with HFpEF.

Udenafil (Zydena), a newly developed PDE-5 inhibitor, has been proved to have similar efficacy and safety profile, compared with other PDE-5 inhibitors. Also, laboratory data showed that udenafil inhibits ventricular hypertrophy and fibrosis in rat heart failure model. Based on these results, we hypothesized that udenafil would improve symptom, exercise capacity and hemodynamic status in patients with HFpEF.

In this 12-week, randomized, double-blind, placebo-controlled trial, patients with HFpEF will be enrolled according to the eligibility criteria. After randomization, study participants will be assigned to receive either 50mg of udenafil or placebo two times a day for 4 weeks, and then the dosage will be doubled to 100mg two times a day for next 8 weeks. Participants will attend study visits at baseline and weeks 4 and 12. Physical examination, medical history review, blood sample collection and electrocardiogram will be conducted on each study visits. At baseline and week 12, participants will undergo cardiopulmonary exercise test and exercise echocardiography. At every study visits, researchers will collect health information.

ELIGIBILITY:
Inclusion Criteria:

* Previous clinical diagnosis of heart failure with preserved ejection fraction (or diastolic heart failure) with current New York Heart association (NYHA) class II-IV symptoms
* Left ventricular ejection fraction (LVEF) greater than or equal to 50%, as determined by echocardiography in the 12 months before study entry
* Has experienced at least one of the following in the 12 months before study entry

  1. Hospitalization for decompensated heart failure
  2. Acute treatment with intravenous loop diuretics or hemofiltration
  3. E/E' ratio greater than or equal to 15 measured by echocardiography
  4. E/E' ratio greater than or equal to 8, and left atrial volume index (LAVI) greater than or equal to 40 ml/m2 measured by echocardiography
  5. E/E' ratio greater than or equal to 8 measured by echocardiography, and plasma BNP concentration greater or equal to 200 pg/ml

Exclusion Criteria:

* History of reduced LVEF (less than 50%)
* Valve disease (greater than mild stenosis or regurgitation)
* Hypertrophic cardiomyopathy
* Infiltrative or inflammatory myocardial disease
* Pericardial disease
* Obstructive or restrictive lung disease
* Primary pulmonary arteriopathy
* Has neuromuscular, orthopedic, or other non-cardiac condition that prevents individual from exercise testing
* Has experienced myocardial infarction or unstable angina, or has undergone percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) within 60 days before study entry
* Non-cardiac illness with estimated life expectancy less than 1 year at the time of study entry, based on the judgment of the physician
* Current use of nitrate therapy
* Current use of other phosphodiesterase 5 inhibitors (ie. sildenafil, vardenafil, tadalafil) for treatment of impotence or pulmonary artery hypertension
* Current use of cytochrome P450 3A4 inhibitors (ie. ketoconazole, itraconazole, erythromycin, saquinavir, cimetidine, protease inhibitors for HIV)
* Severe hypotension (systolic blood pressure [SBP] less than 90mmHg or diastolic blood pressure [DBP] less than 50mmHg) or uncontrolled hypertension (SBP greater than 180mmHg or DBP greater than 100mmHg)
* Resting heart rate (HR) greater than 100bpm
* Known severe renal dysfunction (estimated glomerular filtration rate [GFR] less than 30ml/min/1.73m2 by modified modification of diet in renal disease [MDRD] equation)
* Known severe liver disease (alanine transaminase [ALT] or aspartate aminotransferase [AST] level greater than three times the upper normal limit, alkaline phosphatase [ALP] or total bilirubin greater than two times the upper normal limit)
* History of leukemia, multiple myeloma or penile deformities that increase the risk for priapism (eg. Peyronie's disease)
* History of proliferative diabetic retinopathy, retinitis pigmentosa, nonischemic optic neuropathy, or unexplained visual disturbance
* Female patients currently pregnant or women of childbearing age who were not using contraception
* Listed for heart transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-04 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Change of maximal VO2 in cardiopulmonary exercise test | Baseline and 12th weeks
  Comparison between groups and within groups.

SECONDARY OUTCOMES:
Change of ventilator efficiency (VE/VCO2 slope) in cardiopulmonary exercise test | Baseline and 12th week
  Comparison between groups and within groups.
Change of symptomatic status expressed as New York Heart Association (NYHA) functional class | Baseline, 4th week, and 12th week
  Comparison between groups and within groups.
Change of symptomatic status expressed as Borg dyspnea index | Baseline, 4th week, and 12th week
  Comparison between groups and within groups.
Change of pulmonary artery systolic pressure (PASP) in echocardiography at rest and during exercise | Baseline and 12th week
  Comparison between groups and within groups.
Change of left ventricular systolic function expressed as ejection fraction (EF), fractional shortening (FS) in echocardiography | Baseline and 12th week
  Comparison between groups and within groups.
Change of left ventricular diastolic function expressed as E velocity, E' velocity, E/E' ratio, E/A ratio | Baseline and 12th week
  Comparison between groups and within groups.
Change of left atrial volume | Baseline and 12th week
  Comparison between groups and within groups.
Change of plasma concentration of BNP | Baseline, 4th week, and 12th week
  Comparison between groups and within groups.
All-cause death | 12th week
  The occurrence of all-cause mortality during 12 week follow-up
Cardiac death | 12th week
  The occurrence of cardiac death including sudden cardiac death during 12 week follow-up
Admission for heart failure | 12th week
  Admission due to congestive heart failure during 12 week follow-up
Composite clinical endpoints | 12th week
  Composite clinical endpoints during 12 week follow-up, are defined as follows:
  1. Composite of all-cause death and admission for heart failure
  2. Composite of cardiac death and admission for heart failure
Safety endpoint | 12th week
  Safety endpoint during 12 week follow-up, is defined as follows:
  1. Development of facial flushing, febrile sensation, eyeball pain, visual disturbance, headache, penile erection.
  2. Intolerance or development of other adverse drug reactions related with study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Jin Kim, MD, PhD, Study Chair — Seoul National University Hospital; In-Chang Hwang, MD, Study Director — Seoul National University Hospital; Goo-Yeong Cho, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital; Hyung-Kwan Kim, MD, PhD, Study Director — Seoul National University Hospital; Seung-Pyo Lee, MD, Study Director — Seoul National University Hospital; Kyung-Hee Kim, MD, Study Director — Seoul National University Hospital; Yeonyee E Yoon, MD, Study Director — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Background] Bhatia RS, Tu JV, Lee DS, Austin PC, Fang J, Haouzi A, Gong Y, Liu PP. Outcome of heart failure with preserved ejection fraction in a population-based study. N Engl J Med. 2006 Jul 20;355(3):260-9. doi: 10.1056/NEJMoa051530. PMID 16855266
- [Background] Paulus WJ, Tschope C, Sanderson JE, Rusconi C, Flachskampf FA, Rademakers FE, Marino P, Smiseth OA, De Keulenaer G, Leite-Moreira AF, Borbely A, Edes I, Handoko ML, Heymans S, Pezzali N, Pieske B, Dickstein K, Fraser AG, Brutsaert DL. How to diagnose diastolic heart failure: a consensus statement on the diagnosis of heart failure with normal left ventricular ejection fraction by the Heart Failure and Echocardiography Associations of the European Society of Cardiology. Eur Heart J. 2007 Oct;28(20):2539-50. doi: 10.1093/eurheartj/ehm037. Epub 2007 Apr 11. PMID 17428822
- [Background] Takimoto E, Champion HC, Li M, Belardi D, Ren S, Rodriguez ER, Bedja D, Gabrielson KL, Wang Y, Kass DA. Chronic inhibition of cyclic GMP phosphodiesterase 5A prevents and reverses cardiac hypertrophy. Nat Med. 2005 Feb;11(2):214-22. doi: 10.1038/nm1175. Epub 2005 Jan 23. PMID 15665834
- [Background] Lewis GD, Shah R, Shahzad K, Camuso JM, Pappagianopoulos PP, Hung J, Tawakol A, Gerszten RE, Systrom DM, Bloch KD, Semigran MJ. Sildenafil improves exercise capacity and quality of life in patients with systolic heart failure and secondary pulmonary hypertension. Circulation. 2007 Oct 2;116(14):1555-62. doi: 10.1161/CIRCULATIONAHA.107.716373. Epub 2007 Sep 4. PMID 17785618
- [Background] Guazzi M, Vicenzi M, Arena R, Guazzi MD. PDE5 inhibition with sildenafil improves left ventricular diastolic function, cardiac geometry, and clinical status in patients with stable systolic heart failure: results of a 1-year, prospective, randomized, placebo-controlled study. Circ Heart Fail. 2011 Jan;4(1):8-17. doi: 10.1161/CIRCHEARTFAILURE.110.944694. Epub 2010 Oct 29. PMID 21036891
- [Background] Kim BH, Lim HS, Chung JY, Kim JR, Lim KS, Sohn DR, Cho JY, Yu KS, Shin SG, Paick JS, Jang IJ. Safety, tolerability and pharmacokinetics of udenafil, a novel PDE-5 inhibitor, in healthy young Korean subjects. Br J Clin Pharmacol. 2008 Jun;65(6):848-54. doi: 10.1111/j.1365-2125.2008.03107.x. Epub 2008 Mar 3. PMID 18318773
- [Background] Kang KK, Ahn GJ, Sohn YS, Ahn BO, Kim WB. DA-8159, a new PDE5 inhibitor, attenuates the development of compensatory right ventricular hypertrophy in a rat model of pulmonary hypertension. J Int Med Res. 2003 Nov-Dec;31(6):517-28. doi: 10.1177/147323000303100608. PMID 14708417